CLINICAL TRIAL: NCT00652613
Title: Phase II Study of 3-Dimensional Conformal Radiotherapy (3D-CRT) vs Intensity Modulated Radiotherapy (IMRT) for Squamous Cell Carcinoma of the Head and Neck (HNSCC)
Brief Title: Study of 3-Dimensional Conformal Radiotherapy (3D-CRT) Versus Intensity Modulated Radiotherapy (IMRT) for Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Sarbani Ghosh-Laskar, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H&N_3DCRT_IMRT07
Record Dates: First submitted 2008-03-27; First posted 2008-04-04 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: 3DCRT; IMRT; HNSCC; Quality of life; Major salivary gland sparing; Pattern of local and loco-regional recurrence; Disease Free Survival (DFS) & Overall Survival (OAS); Dose reduction to normal structures with IMRT
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 3 dimensional conformal radiotherapy
  Interventions: Radiation: 3 Dimensional Radiation Therapy
- 2 (Experimental): Intensity Modulated Radiation Therapy (IMRT)
  Interventions: Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Radiation: 3 Dimensional Radiation Therapy — Radiation with 6 MV photons to dose of 70Gy/ 35#/ 7 weeks
  Arms: 1
Radiation: Intensity Modulated Radiation Therapy — IMRT with 6 MV photons to a dose of 66Gy/30#/ 6 weeks
  Arms: 2

SUMMARY:
Head & Neck squamous cell carcinomas are the commonest cancers afflicting the developing countries. Traditionally surgery or radiotherapy alone in the early stages and surgery with postoperative radiotherapy in advanced stages have been the mainstay of treatment. Of late there has been a paradigm shift in the management of these cancers, particularly those of the oropharynx and laryngopharynx, where chemoradiation has been advocated as part of organ preservation protocol with good outcomes. Conventional radiotherapy involves the use of 2 or 3 field technique with or without compensators to encompass the volume at risk to radical doses of 66-70 Gy typically needed to sterilize gross disease. This strategy however is associated with considerable acute morbidity (mucositis, dysphagia, dermatitis) and debilitating late toxicity (xerostomia). Three dimensional conformal radiation therapy (3D-CRT) and intensity modulated radiation therapy (IMRT) have the potential to improve the dose distribution, with increased doses to the target volumes and reduced doses to surrounding normal structures, thereby improving the therapeutic ratio.

DETAILED DESCRIPTION:
1.0 Introduction: Head & Neck squamous cell carcinomas are the commonest cancers afflicting the developing countries. Traditionally surgery or radiotherapy alone in the early stages and surgery with postoperative radiotherapy in advanced stages have been the mainstay of treatment. Of late there has been a paradigm shift in the management of these cancers, particularly those of the oropharynx and laryngopharynx, where chemoradiation has been advocated as part of organ preservation protocol with good outcomes. Conventional radiotherapy involves the use of 2 or 3 field technique with or without compensators to encompass the volume at risk to radical doses of 66-70 Gy typically needed to sterilize gross disease. This strategy however is associated with considerable acute morbidity (mucositis, dysphagia, dermatitis) and debilitating late toxicity (xerostomia). Three dimensional conformal radiation therapy (3D-CRT) and intensity modulated radiation therapy (IMRT) have the potential to improve the dose distribution, with increased doses to the target volumes and reduced doses to surrounding normal structures, thereby improving the therapeutic ratio.

2.0 Objectives: 2.1 To compare the major salivary gland sparing by 3-D CRT vis-à-vis IMRT and assess the adequacy of target volume coverage with these conformal techniques.

2.2 To determine the pattern of local and loco-regional recurrence. 2.3 To determine Disease Free Survival (DFS) & Overall Survival (OAS) 2.4 To study the quality of life of these patients 2.5 To assess the reduction in dose with IMRT to the normal larynx & normal pharyngeal constrictors in oropharyngeal cancers, uninvolved oral mucosa and middle & inner ear apparatus in both oropharyngeal & laryngopharyngeal cancers

3.0 Patient Selection: 3.1 Eligibility 3.1.1 Biopsy proven squamous cell carcinoma of the oropharynx or laryngopharynx.

3.1.2. AJCC stage T1-3, NO-2b, MO patients with pre-treatment tumor measurements clinically as well as on CT/MRI scans. 3.1.3 Surgery of the primary tumor limited to excisional or incisional biopsy. 3.1.4 No form of neck dissection for nodal metastases. 3.1.5 KPS > 60 (see appendix I). 3.1.6 Age > 18 and < 65 years. 3.1.7 No prior history of therapeutic irradiation. 3.1.8 Patient willing and reliable for follow-up. 3.1.9 Patient's nutritional & physical condition compatible with planned therapy.

3.1.10 Signed study specific consent form (see Appendix II). 3.2 Ineligibility criteria: 3.2.1 Evidence of distant metastases. 3.2.2 Previous therapeutic irradiation for head & neck cancer or any other invasive cancer other than squamous or basal cell carcinoma of the skin. 3.2.3 History of prior malignancy. 3.2.4 Prophylactic use of amifostine or pilocarpine. 3.2.5 Active untreated infection like tuberculosis, which preclude the use of systemic chemotherapy or would interfere with completion of treatment. 3.2.6 Any histopathology other than Squamous Carcinoma. 3.2.7 Primary nasopharyngeal carcinoma. 3.2.8 Age < 18 or > 65 years. 3.2.9 Pregnancy or lactating women. 4.0 Pre-treatment evaluation: 4.1 All patients required to complete the following prior to start of therapy: 4.1.1 Complete history and physical examination including weight and height. 4.1.2. Complete diagrammatic and descriptive documentation of the extent of disease, both primary and regional following appropriate endoscopic procedures. 4.1.3 Complete dental and nutritional evaluation. All dental repair to be done at least one week prior to starting therapy. 4.1.4 Completion of the following laboratory investigations: CBC, LFT, RFT, TFT, baseline speech assessment and audiometric assessment. 4.1.5 Completion of the following radiological investigations: CXR, CT/MRI of the head & neck with volumetric assessments, Planning scan with contrast (unless otherwise contraindicated) with 3mm contiguous slices in appropriate immobilization systems. A PET scan or a CT-PET hybrid scan may be done at the discretion of the treating physician (Appendix III). Bone scan and liver scan as per clinical indication.

4.1.6 Salivary scintigraphy for the parotid glands. 4.1.7 A baseline QOL questionnaire (Appendix IV) will be filled in for each patient.

5.0 Radiation therapy: 5.1 Treatment planning, imaging & localization requirements. 5.1.1 Immobilization: In supine position with a customized thermoplastic device.

5.1.2 Planning scan: Contrast enhanced planning CT scan of the area of interest with 3mm slices on CT-simulator that is networked to the treatment planning system (Cadplan).

5.1.3 Target delineation: Planning target volumes (GTV and CTV) and organ at risk volumes (spinal cord and both the parotids) to be contoured on each slice. Other organs such as uninvolved oral mucosa, middle & inner ear and normal larynx & pharyngeal constrictors in oropharyngeal cancers also to be contoured on each slice. An isometric margin of 5mm to be provided to the CTV for final PTV and 3mm to organs at risk for planning organ at risk volume (PORV). The GTV will include only the primary and involved neck nodes. The delineation of the various volumes will be as per consensus guidelines. The priorities and constraints for IMRT plan will also be decided on a case to case basis (see appendix V for details).

5.1.4 Prescription: The goal of the treatment plan would be to encompass the PTV subclinical disease with a dose of 60-54 Gy conventional fractionation equivalent and the GTV with 70 Gy equivalent while sparing as much of the aforesaid critical structures as possible without compromising on the GTV. Primary target (gross disease with margins) dose will be 70 Gy conventional fractionation equivalent (70 Gy/35#/7 weeks with 3-D CRT ad 66 Gy/30#/6 weeks with IMRT). The secondary target (sub-clinical disease) dose will be 50-54 Gy conventional fractionation equivalent (50-54 Gy/28-30#/5.5-6 weeks with 3-D CRT and 54 Gy/30#/6 weeks with IMRT). An optional secondary target area may be defines as area of high risk disease (e.g. first echelon nodes). This shall receive 60 Gy/30#/6 weeks with both 3-D CRT and IMRT.

The maximum permissible point doses to the spinal cord will be limited to 40 Gy. All patients to be planned with both 3-D CRT as well as IMRT, irrespective of the final treatment protocol. 3-D CRT planning to be done on Cadplan/Eclipse (Varian, USA) using multileaf collimators (MLCs) for beam shaping. IMRT planning to be done using Helios inverse planning module of Cadplan/Eclipse. Treatment to be delivered on a Varian LINAC (2100 CD or 6 Ex) using dynamic MLCs (sliding window technique).

5.1.5 Plan evaluation: Comparative evaluation of the bease 3-D CRT and IMRT plan for the individual patient to be done. Cumulative dose volume histograms (DVHs) to be computed for PTV and each PORV to assist in plan evaluation. Plans to be compared with respect to conformal avoidance of organs at risk, conformity index, homogeneity index and DVHs. An in detail evaluation of the quality assurance (Appendix VI) and dosimetric methods involved in the procedure would also be carried out and will be correlated with final outcome.

6.0 Other therapy: 6.1 Chemotherapy: Concurrent platinum based chemotherapy to be considered for all patients with T3 or N+ disease.

6.2 Cytoprotectors: Use of amifostine or pilocarpine is not allowed. 7.0 Patient assessments: 7.1 Patients assessments table (see Appendix VII for details). 7.2 Evaluation 7.2.1 Every follow up visit: All patients require to follow up 6weeks and 12 weeks from end of radiotherapy, Thereafter follow up visits would be scheduled three monthly for the first two years and annually thereafter. Routine head & neck examination, including endoscopic examination will be performed at the first follow-up and thereafter as and when needed, performance status, weight, toxicity and QOL documentation will be carried out at each follow-up. Salivary scintigraphy, swallowing status, speech assessment, thyroid function test and audiometry will be done at first follow-up post treatment and six monthly thereafter. Follow-up PET scan to be done at the discretion of the treating physician. Dental care to be provided as and when needed.

7.2.2 Other studies: CXR for persistent cough, hemoptysis or chest pain; skeletal survey or bone scan in case of any bone pains and biopsy of any suspicious lesion in the upper aero-digestive tract.

7.2.3 Objective response criteria (see Appendix VIII). 7.3 Criteria for removal from treatment 7.3.1 Progression of disease while on treatment 7.3.2 Withdrawal of consent by patient 7.3.3 Severe radiation morbidity resulting in a break of 2 weeks or more. 8.0 Data Collection: 8.1 Summary of data submission ITEM DUE Demographic form Within 2 weeks of study entry Initial Evaluation form 1 week before RT start Diagnostic Pathology Report Before RT start Baseline QOL assessment 1 week before start of treatment Radiotherapy form Within 1 week of end of RT Adverse Event form (see appendix IX for details) Initial follow-up form At 6 weeks from end of RT Follow-up forms At 3, 6 & 12 Months from end of RT Long term follow-up forms Yearly after 5 years Autopsy report If needed

8.2 Summary of RT QA requirements (see Appendix VI for details): Preliminary Dosimetric Information Within 1 week of start of RT Simulation & Port films Every week Final Dosimetric Information Within 1 week of end of RT

Hard copy of isodoses and DVH for total plan including any charges

9.0 Statistical consideration: 9.1.1 The primary end point is acute salivary gland toxicity (> = Gr 2) as per the RTOG toxicity criteria (see Appendix X & XI). This is also to be assessed by salivary scintigraphy and subjectively by patient self-assessment. As a surrogate dose volume histogram shall be used for assessment for major salivary gland sparing.

9.1.2 Secondary endpoints include: a) Local & Loco-regional control b) DFS & c) OAS 9.2 Patient accrual, sample size & analysis: 60 patients. 9.2.1 Approximately 85% of patients with conventional techniques or 3-D CRT would develop acute salivary gland toxicity of grade 2 or more. With IMRT, it is hypothesized that this could be reduced to 50%. The total number of patients needed would be fifty-four assuming alpha error 0.05 and beta error 0.20 (one tailed test). The projected 3 year locoregional control rate for this group is 70%. Ensuring that the salivary gland sparing should not be at the expense of loco-regional control, the upper limit for locoregional failure rate is set at 45% as per Fleming's one step multiple testing procedure. In case this is exceeded anytime during the interim analysis, the entire protocol shall be re-examined.

9.2.2 Sixty patients to be accrued over a 24 month period from date of start 9.2.3 Interim analysis of toxicity and accrual data planned every six months. Initial results of treatment to be reported when all patients have completed at least 6 months on follow-up. Final results to be reported at a minimum of 2 year follow-up on all patients.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven squamous cell carcinoma of the oropharynx or laryngopharynx.
* AJCC stage T1-3, NO-2b, MO patients with pre-treatment tumor measurements clinically as well as on CT/MRI scans.
* Surgery of the primary tumor limited to excisional or incisional biopsy.
* No form of neck dissection for nodal metastases.
* KPS > 60 (see appendix I).
* Age > 18 and < 65 years.
* No prior history of therapeutic irradiation.
* Patient willing and reliable for follow-up.
* Patient's nutritional & physical condition compatible with planned therapy.

Exclusion Criteria:

* Evidence of distant metastases.
* Previous therapeutic irradiation for head & neck cancer or any other invasive cancer other than squamous or basal cell carcinoma of the skin.
* History of prior malignancy.
* Prophylactic use of amifostine or pilocarpine.
* Active untreated infection like tuberculosis, which preclude the use of systemic chemotherapy or would interfere with completion of treatment.
* Any histopathology other than Squamous Carcinoma.
* Primary nasopharyngeal carcinoma.
* Age < 18 or > 65 years.
* Pregnancy or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Major salivary gland sparing by 3-D CRT vis-à-vis IMRT. Assess adequacy of target volume coverage | 4 yrs
Determine the pattern of local and loco-regional recurrence | 4 yrs

SECONDARY OUTCOMES:
Disease Free Survival (DFS) and Overall Survival (OAS) | 4 yrs
Quality of life 3. Dose to OAR | 4 yrs
Assess the reduction in dose with IMRT to the normal larynx and normal pharyngeal constrictors in oropharyngeal cancers, uninvolved oral mucosa and auditory apparatus | 4 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Sarbani Ghosh-Laskar, MD, Principal Investigator — Department of Radiation Oncology, Tata Memorial Centre; Ketayun Dinshaw, FRCR, Study Director — Director, Tata Memorial Centre
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- [Derived] Ghosh-Laskar S, Yathiraj PH, Dutta D, Rangarajan V, Purandare N, Gupta T, Budrukkar A, Murthy V, Kannan S, Agarwal JP. Prospective randomized controlled trial to compare 3-dimensional conformal radiotherapy to intensity-modulated radiotherapy in head and neck squamous cell carcinoma: Long-term results. Head Neck. 2016 Apr;38 Suppl 1:E1481-7. doi: 10.1002/hed.24263. Epub 2015 Nov 11. PMID 26561342